CLINICAL TRIAL: NCT05011513
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 2/3, DOUBLE-BLIND, 2 ARM STUDY TO INVESTIGATE ORALLY ADMINISTERED PF 07321332/RITONAVIR COMPARED WITH PLACEBO IN NONHOSPITALIZED SYMPTOMATIC ADULT PARTICIPANTS WITH COVID-19 WHO ARE AT LOW RISK OF PROGRESSING TO SEVERE ILLNESS
Brief Title: Evaluation of Protease Inhibition for COVID-19 in Standard-Risk Patients (EPIC-SR).
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Enrollment ceased due to a very low rate of hospitalization or death observed in the standard-risk patient population
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4671002; 2021-002857-28 (EudraCT Number); EPIC-SR (Other: Alias Study Number)
Record Dates: First submitted 2021-07-30; First posted 2021-08-18 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Intervention Model Description: Eligible participants with a confirmed diagnosis of SARS-CoV-2 infection will be randomized (1:1) to receive PF-07321332/ritonavir or placebo orally every 12 hours for 5 days (10 doses total).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07321332/ritonavir (Experimental): Orally administered PF-07321332+ritonavir
  Interventions: Drug: PF-07321332; Drug: Ritonavir
- Placebo (Placebo Comparator): Orally administered Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07321332 — PF-07321332 (tablet)
  Arms: PF-07321332/ritonavir
Drug: Ritonavir — Ritonavir (capsule)
  Arms: PF-07321332/ritonavir
Drug: Placebo — Placebo (tablet)
  Arms: Placebo
Drug: Placebo — Placebo (capsule)
  Arms: Placebo

SUMMARY:
The primary hypothesis to be tested is whether or not there is a difference in time to sustained alleviation of all targeted COVID-19 signs and symptoms through Day 28 between PF-07321332/ritonavir and placebo.

DETAILED DESCRIPTION:
Throughout the study period, provision will be made to allow study visits to be conducted at a participant's home or at another non-clinic location, if available. The total study duration is up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection 5 days prior to randomization
* Initial onset of COVID-19 signs/symptoms within 5 days of randomization
* Fertile participants must agree to use a highly effective method of contraception

Exclusion Criteria:

* Has at least one underlying medical condition associated with an increased risk of developing severe illness from COVID-19
* History of or need for hospitalization for the medical treatment of COVID-19
* Prior diagnosis of SARS-CoV-2 infection (reinfection)
* Known medical history of liver disease
* Receiving dialysis or have known renal impairment
* Known Human Immunodeficiency Virus (HIV) infection with viral load > 400 copies/ml or taking prohibited medications for HIV treatment
* Suspected or confirmed concurrent active systemic infection other than COVID-19
* Current or expected use of any medications or substances that are highly dependent on Cytochrome P450 3A4 (CYP3A4) for clearance or are strong inducers of CYP3A4
* Has received or is expected to receive monoclonal antibody treatment or convalescent COVID-19 plasma
* Has received any SARS-CoV-2 vaccine within 12 months of screening
* Participating in another interventional clinical study with an investigational compound or device, including those for COVID-19
* Known prior participation in this trial or other trial involving PF-07321332
* Oxygen saturation of < 92% on room air
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (225):
- United States (78):
  - Cahaba Research Inc, Pelham, Alabama
  - The Institute for Liver Health dba Arizona Clinical Trials, Mesa, Arizona
  - Matrix Mobile Health Clinic #49, #35, and #62, Scottsdale, Arizona
  - The Institute for Liver Health dba Arizona Clinical Trials, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Lightship, El Segundo, California
  - Ascada Research, Fullerton, California
  - Atella Clinical Research LLC., La Palma, California
  - Ark Clinical Research, Long Beach, California
  - South Bay Clinical Research Institute, Redondo Beach, California
  - Benchmark Research, Sacramento, California
  - Optimus Medical Group, San Francisco, California
  - Hope Clinical Research (COVID Satellite Site), West Hills, California
  - Future Innovative Treatments, LLC, Colorado Springs, Colorado
  - Synergy Healthcare, Bradenton, Florida
  - MOORE Clinical Research, Inc., Brandon, Florida
  - TrueBlue Clinical Research, Brandon, Florida
  - Herco Medical and Research Center Inc, Coral Gables, Florida
  - Advance Clinical Research Group, Cutler Bay, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Omega Research Orlando, LLC, DeBary, Florida
  - Eastern Research Inc, Hialeah, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Doral Medical Research, LLC, Hialeah, Florida
  - Unlimited Medical Research Group, LLC, Hialeah Gardens, Florida
  - ASCLEPES Research Centers, Lutz, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Premium Medical Research Corp, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - I.V.A.M. Clinical & Investigational Center, LLC, Miami, Florida
  - C'A Research, Miami, Florida
  - ProLive Medical Research, Corp., Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Clinical Site Partners, Inc d/b/a CSP Miami, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Pro-Care Research Center, Corp., Miami Gardens, Florida
  - Savin Medical Group, LLC, Miami Lakes, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - CDC Research Institute, Port Saint Lucie, Florida
  - USPA Advance Concept Medical Research Group LLC, South Miami, Florida
  - ASCLEPES Research Centers, Spring Hill, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Clinical Site Partners, Inc. dba CSP Orlando, Winter Park, Florida
  - Accellacare, Ames, Iowa
  - McFarland Clinic, PC, Ames, Iowa
  - New Orleans Sinus Center (COVID-19 Testing), Marrero, Louisiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Southern Clinical Research Associates, LLC, Metairie, Louisiana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Excel Clinical research, Las Vegas, Nevada
  - AXCES Research Group, Santa Fe, New Mexico
  - NYC Health + Hospitals / Harlem, New York, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Innovo Research: Wilmington Health, Wilmington, North Carolina
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - Avera Research Institute, Sioux Falls, South Dakota
  - PharmaTex Research, LLC, Amarillo, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - St Hope Foundation, Bellaire, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - SignatureCare Emergency Center, Houston, Texas
  - Trio Clinical Trials, LLC, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Epic Medical Research, Red Oak, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - BFHC Research, San Antonio, Texas
  - Tranquility Research, Webster, Texas
  - TMPG Clinical Research, Newport News, Virginia
  - TPMG Clinical Research, Newport News, Virginia
- Argentina (5):
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Instituto Médico de la Fundación Estudios Clínicos (Fundación Estudios Clínicos), Rosario, Santa Fe Province
  - Hospital de Clinicas Presidente Nicolas Avellaneda, San Miguel de Tucumán, Tucumán Province
  - Clinica Mayo Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Centro Médico de Córdoba, Córdoba
- Brazil (15):
  - Chronos Pesquisa Clinica, Brasília, Federal District
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas - INI/FIOCRUZ, Rio de Janeiro, Rio de Janeiro
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas, Natal, Rio Grande do Norte
  - Hospital De Clinicas De Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CECOR - Centro Oncológico de Roraima, Boa Vista, Roraima/rr
  - Hospital Dia do Pulmao, Blumenau, Santa Catarina
  - Hospital e Maternidade Celso Pierro - PUC Campinas / Sociedade Campineira de Educação e Instruçã, Campinas, São Paulo
  - CECIP JAÚ - Centro de Estudos Clínicos do Interior Paulista - LTDA, Jaú, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Unidade Referenciada Oswaldo Cruz Vergueiro, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, São Paulo
  - Instituto de Infectologia Emilio Ribas, São Paulo
- Bulgaria (23):
  - Individual Practice for Primary Medical Care - IPPMC - Dr. P. Panayotov EOOD, Burgas
  - "Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases-Haskovo" Ltd, Haskovo
  - MHAT "Sv.Ivan. Rilski'' Kozloduy EOOD, Kozloduy
  - Diagnostic-Consultative Center I Lom EOOD, Lom
  - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz EOOD, Lom
  - Medical centre Leo Clinic EOOD, Lovech
  - MHAT Heart and Brain EAD, Pleven
  - DCC Sveti Georgi EOOD, Plovdiv
  - MHAT "St. Panteleimon "- Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveti Ivan Rilski - Razgrad AD, Razgrad
  - "Specialized Hospital for Active Treatment of Pneumo-Physiatric Diseases Dr. Dimitar Gramatikov -, Rousse
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Samokov
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Multiprofile hospital for active treatment - Sliven to Military Medical Academy, Sliven
  - Diagnostic-Consultative Center XXII- Sofia ЕООD, Sofia
  - UMHATEM N. I. Pirogov EAD, Sofia
  - MHAT "St. Sofia" EOOD, Sofia
  - Specialized hospital for active treatment in pulmonology and phthisiology "Stara Zagora" EOOD, Stara Zagora
  - Multiprofile Hospital for Active Treatment Targovishte AD, Targovishte
  - Outpatient Clinic for Primary Outpatient Medical Care "Puls" - Dr. Mladen Buchvarov EOOD, Tsarevo
  - Medical center Leo Clinic EOOD, Varna
  - MOBAL "D-r Stefan Cherkezov" AD, Veliko Tarnovo
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases Vratsa EOOD, Vratsa
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica CIC, Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, CIREEM S.A.S, Bogota, Cundinamarca
  - Fundacion Cardiomet Cequin, Armenia, Quindío Department
- Czechia (2):
  - Zdraví-Fit, s.r.o., Protivín
  - Nemocnice Slany, Slaný
- Hungary (7):
  - Trial Pharma Kft., Békéscsaba
  - Semmelweis University Varosmajori Sziv Es Ergyogyaszati Klinika, Budapest
  - Varosmajori Sziv- es Ergyogyaszati Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont Infektologiai Klinika, Debrecen
  - Agria-Study Kft., Eger
  - Trial Pharma Kft., Gyula
  - Medifarma-98 Kft., Nyíregyháza
- Japan (5):
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Tokyo Shinagawa Hospital, Shinagawa-ku, Tokyo
  - Sekino Hospital, Toshimaku, Tokyo
  - Kyushu Medical Center, Fukuoka
- Malaysia (4):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Taiping, Taiping, Perak
  - Hospital Miri, Miri, Sarawak
  - Klinik Kesihatan Kuang, Rawang, Selangor
- Mexico (11):
  - Clinical Research Institute S.C., Saltillo, Coahuila
  - Asociación Mexicana para la Investigación Clínica A.C., Pachuca, Hidalgo
  - JM Research SC, Cuernavaca, Morelos
  - Christus - Latam Hub Center of Excellence and Innovation Center S.C., Monterrey, Nuevo León
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - EME RED Hospitalaria, Mérida, Yucatán
  - Kohler & Milstein Research S.A. De C.V., Mérida, Yucatán
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - FAICIC Clinical Research, Veracruz
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- Poland (4):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Badań Klinicznych Piotr Napora Lekarze Spółka Partnerska, Wroclaw
- Puerto Rico (2):
  - Clinical Research Management Group Inc, Ponce
  - Advance Medical Research Center, San Juan
- Delta Health Care srl, Bucharest, Romania
- Slovakia (4):
  - HODOSI - MED, s.r.o., Moldava nad Bodvou
  - MUDr. Viliam Cibik, PhD., s.r.o., Pruské
  - Plucna ambulancia Hrebenar, s.r.o., Spišská Nová Ves
  - ALERGIA s.r.o., Topoľčany
- South Africa (13):
  - Global Clinical Trials, Port Elizabeth, Eastern Cape
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Reimed Vosloorus, Boksburg, Gauteng
  - Lenasia Clinical Trial Centre, Johannesburg, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Clinical Trial Systems (Pty) Ltd, Pretoria, Gauteng
  - Sandton Medical Clinic, Sandton, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - Synapta Clinical Research Center, Durban, KwaZulu-Natal
  - Dr PJ Sebastian Clinical Research Centre, Durban, KwaZulu-Natal
  - Ahmed Al-Kadi Private Hospital, Mayville, Durban, KwaZulu-Natal
  - TASK Eden, George, Western Cape
  - Be Part Research Pty (Ltd), Paarl, Western Cape
- South Korea (3):
  - Chonnam National University Bitgoeul Hospital, Gwangju
  - Boramae Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (7):
  - Eba Centelles, Centelles, Barcelona [barcelona]
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - IMED Valencia, Burjassot, Valencia
  - Complexo Hospitalario Universitario da Coruna, A Coruña
  - Hospital Universitario de la Paz, Madrid
  - Hospital Universitario Virgen de Valme, Seville
- Thailand (9):
  - Bangkok Centre Hotel, Bang Rak, Bangkok
  - Siriraj Hospital, Mahidol University, BangkokNoi, Bangkok
  - Riverside Bangkok Hotel, Bangplud, Bangkok
  - Thai Red Cross Emerging Infectious Diseases (EDI) Clinic, Pathumwan,, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),, Pathumwan, Bangkok
  - Baiyoke Suite Hotel, Ratchathewi, Bangkok
  - Department of Internal Medicine, Faculty of Medicine, Prince of Songkla University,, Hat Yai, Changwat Songkhla
  - Khon Kaen Univerisity Field Hospital, Student Dormitory 26, Khon Kaen University, Khon Kaen
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (15):
  - Cukurova University Medical Faculty, Balcali, Adana
  - Ankara University Medical Faculty, Ibni-Sina Hospital, Ankara
  - Hacettepe University Medical Faculty Hospital, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Uygulama ve Arastirma Hastanesi, Gaziantep
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa-Cerrahpasa Medical Faculty, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - Acibadem University Atakent Hospital, Istanbul
  - Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul
  - Izmir Suat Seren Chest Disease and Surgery Training and Research Hospital, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Mersin University Medical Faculty, Mersin
  - Sakarya University Training and Research Hospital, Sakarya
  - Karadeniz Teknik Universitesi Farabi Hastanesi, Trabzon
- Ukraine (14):
  - Regional Communal Nonprofit Institution "Chernivtsi Regional Clinical Hospital", Chernivtsi
  - Communal non-commercial Enterprise "City Clinical Hospital №3" of Chernivtsi City Council, Chernivtsi
  - Municipal Nonprofit Enterprise "Ivano-Frankivsk Regional Clinical Infectious Diseases Hospital of, Ivano-Frankivsk
  - Municipal Non-profit Enterprise "Ivano-Frankivsk Regional Phthisiopulmonology Center of, Ivano-Frankivsk
  - Communal nonprofit enterprise "Central City Clinical Hospital of Ivano-Frankivsk City Council", Ivano-Frankivsk
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council "Regional Clinical Infectious Diseases, Kharkiv
  - Municipal Non-profit Enterprise "Oleksandrivska Kyiv City Clinical Hospital" Of Executive Body Of, Kyiv
  - Municipal non-commercial enterprise "Kyiv City Clinical Hospital #1" Of Executive Body Of the Kyiv, Kyiv
  - Kyiv Railway Clinical Hospital No.2 of Branch "Health Center of the Public Joint Stock Company, Kyiv
  - Polyclinic of Center for Medical Services and Rehabilitation of State Joint-Stock Holding Company, Kyiv
  - Municipal Nonprofit Enterprise "Lviv City Clinic Hospital #4", Lviv
  - Municipal Enterprise "Poltava Regional Clinical Infectious Diseases Hospital" of Poltava Regional, Poltava
  - Municipal Non-commercial Enterprise "Vinnytsia City Clinical Hospital №1", Vinnytsia
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown TM, Kanu C, Harrington M. Assessing participants' experiences with the COVID-19 symptom diary in a clinical trial. J Patient Rep Outcomes. 2025 Aug 11;9(1):99. doi: 10.1186/s41687-025-00901-5. PMID 40788441
- [Derived] Baniecki ML, Guan S, Rai DK, Yang Q, Lee JT, Hao L, Weinstein E, Hyde C, Cardin RD, Soares H, Hammond J. Integrated virologic analysis of resistance to nirmatrelvir/ritonavir in individuals across four phase 2/3 clinical studies for the treatment of COVID-19. EBioMedicine. 2025 Aug;118:105819. doi: 10.1016/j.ebiom.2025.105819. Epub 2025 Jun 30. PMID 40592258
- [Derived] Hammond J, Fountaine RJ, Yunis C, Fleishaker D, Almas M, Bao W, Wisemandle W, Baniecki ML, Hendrick VM, Kalfov V, Simon-Campos JA, Pypstra R, Rusnak JM. Nirmatrelvir for Vaccinated or Unvaccinated Adult Outpatients with Covid-19. N Engl J Med. 2024 Apr 4;390(13):1186-1195. doi: 10.1056/NEJMoa2309003. PMID 38598573
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as determined by reverse transcription polymerase chain reaction (RT-PCR) within 5 days prior to randomization were included in the study.
Pre-assignment Details: A total of 1440 participants signed informed consent form. Out of which, 1296 subjects were randomized and assigned to study drug. 1288 participants were treated and remaining 8 participants were not treated.
Groups:
- Nirmatrelvir 300 Milligram (mg) + Ritonavir 100 mg: Participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally every 12 hours from Day 1 to 5
- Placebo: Participants were randomized to receive placebo matched to nirmatrelvir/ritonavir every 12 hours for 10 doses from Day 1 through Day 5.
Period: Overall Study
Arm/Group | Nirmatrelvir 300 Milligram (mg) + Ritonavir 100 mg | Placebo
Started | 658 | 638
Treated | 654 | 634
Completed | 632 | 618
Not Completed | 26 | 20
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received. A randomized but not treated participant was excluded from the safety analyses.
Groups:
- Nirmatrelvir 300 mg + Ritonavir 100 mg: Participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally every 12 hours from Day 1 to 5.
- Total: Total of all reporting groups
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo | Total
Number analyzed (Participants) | 654 | 634 | 1288
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.76 (13.47) | 42.63 (13.13) | 42.18 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344 | 352 | 696
  Male | 310 | 282 | 592
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 272 | 261 | 533
  Not Hispanic or Latino | 378 | 367 | 745
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 39 | 32 | 71
  Asian | 69 | 72 | 141
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 23 | 51
  White | 512 | 498 | 1010
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Alleviation of Overall COVID-19 Signs and Symptoms Through Day 28
Description: Sustained alleviation of targeted COVID-19 signs/symptoms was defined as the event occurring on the first 4 consecutive days when all symptoms scored as moderate or severe at the time of enrollment were scored as mild or absent and those scored mild or absent at the time of enrollment were scored as absent. Missing severity at baseline was considered as mild. Time to sustained alleviation of all targeted COVID-19 signs and symptoms through Day 28, was calculated as time (days) from start of study intervention or placebo (Day 1) until sustained alleviation of all targeted COVID-19 associated signs and symptoms. In this outcome measure time to sustained alleviation is reported consolidated for overall COVID-19 signs and symptoms.
Time Frame: From Day 1 to Day 28
Population: Modified intent-to-treat (mITT1) population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Days | 12.000 [11.000 to 13.000] | 13.000 [12.000 to 14.000]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.6027, Log Rank

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious AEs and AEs Leading to Study and Study Drug Discontinuation
Description: An AE was defined as any untoward medical occurrence in a participant or clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening ; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity ; congenital anomaly/birth defect; or that was considered as an important medical event. TEAEs were defined as events that started on or after the study medication start date and time. AEs included both serious and all non-serious adverse events. AEs that led to study discontinuation and AEs that led to discontinuation of study intervention and then continued study were also reported in this outcome measure.
Time Frame: From start of study intervention (Day 1) up to Day 34
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Participants
  TEAEs | 169 | 153
  SAEs | 8 | 13
  AEs led to discontinuation of study | 0 | 1
  AEs led to discontinue study intervention and continued study | 16 | 5

3. Secondary Outcome: Percentage of Participants With COVID-19 Related Hospitalization or Death From Any Cause Through Day 28
Description: Percentage of participants with COVID-19 related hospitalization or death from any cause during the first 28 days of the study was estimated using the Kaplan-Meier (KM) method.
Time Frame: From Day 1 to Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Percentage of participants
  COVID-19 hospitalization | 0.765 | 1.577
  Death | 0 | 0.158
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.1796, Normal approximation — P-value reported for COVID-19 hospitalization and death due to any cause

4. Secondary Outcome: Percentage of Participants With Death Through Week 24
Description: Percentage of participants with death (all-cause) event were reported in this outcome measure.
Time Frame: From Day 1 to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Percentage of participants | 0 | 0.2

5. Secondary Outcome: Number of COVID-19 Related Medical Visits Per Day Through Day 28
Description: Number of COVID-19 related medical visits per day were reported in this outcome measure.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Medical visits per day
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Medical visits per day | 0.0010 [0.0005 to 0.0019] | 0.0020 [0.0010 to 0.0038]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.0971, Negative binomial

6. Secondary Outcome: Duration of Hospitalization and Intensive Care Unit (ICU) Stay Through Day 28
Time Frame: From Day 1 to Day 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Days
  Hospitalization | 0.049 (0.591) | 0.181 (1.787)
  ICU | 0.000 (0.000) | 0.065 (1.004)

7. Secondary Outcome: Percentage of Participants With Severe Signs and Symptoms of COVID-19 Through Day 28
Description: Participants recorded a daily severity rating of their symptom severity over the past 24 hours based on a 4-point scale in which 0 was reported if no symptoms were present; 1 if mild; 2 if moderate; and 3 if severe. A participant with severe score for any targeted symptoms post-baseline was counted as severe. Vomiting and diarrhea each was rated on a 4-point frequency scale where 0 was reported for no occurrence, 1 for 1 to 2 times, 2 for 3 to 4 times, and 3 for 5 or greater. Sense of smell and sense of taste each be rated on a 3-point Likert scale where 0 was reported if the sense of smell/taste was the same as usual, 1 if the sense of smell/taste was less than usual, and 2 for no sense of smell/taste.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 648 | 633
Percentage of participants | 19.136 | 21.643
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Main effects of treatment, geographic region, baseline SARS-CoV-2 serology status and baseline viral load (< 4 log10 copies/mL, >= 4 log10 copies/mL); Test type: Superiority; p = 0.1622, Regression, Logistic; Odds Ratio (OR) = 0.819, 95% CI 2-sided [0.618 to 1.084]

8. Secondary Outcome: Time to Sustained Resolution of Overall COVID-19 Signs and Symptoms Through Day 28
Description: Sustained resolution was defined as when targeted symptoms are scored as absent for 4 consecutive days. The first day of the 4 consecutive-day period was considered the first event date.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized. In this outcome measure time to sustained resolution is reported consolidated for overall COVID-19 signs and symptoms. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 428 | 425
Days | 15.000 [14.000 to 16.000] | 16.000 [15.000 to 17.000]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.4298, Log Rank

9. Secondary Outcome: Time to Sustained Alleviation of Each COVID-19 Signs and Symptoms Through Day 28
Description: Sustained alleviation of targeted COVID-19 signs/symptoms was defined as the event occurring on the first 4 consecutive days when all symptoms scored as moderate or severe at the time of enrollment were scored as mild or absent and those scored mild or absent at the time of enrollment were scored as absent. Missing severity at baseline was treated as mild. Time to sustained alleviation of all targeted COVID-19 signs and symptoms through Day 28, was calculated as time (days) from start of study intervention or placebo (Day 1) until sustained alleviation of all targeted COVID-19 associated signs and symptoms. In this outcome measure time to sustained alleviation is reported for each COVID-19 signs and symptoms.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized. Here, ''Number Analyzed'' signifies participants evaluable at specific rows.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Days
  Muscle or body aches: number analyzed (Participants) | 466 | 449
  Muscle or body aches | 5.000 [4.000 to 6.000] | 5.000 [4.000 to 6.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 222 | 205
  Shortness of breath or difficulty breathing | 5.000 [4.000 to 6.000] | 6.000 [5.000 to 7.000]
  Chills or shivering: number analyzed (Participants) | 318 | 319
  Chills or shivering | 3.000 [3.000 to 4.000] | 3.000 [3.000 to 4.000]
  Cough: number analyzed (Participants) | 512 | 502
  Cough | 7.000 [6.000 to 8.000] | 8.000 [7.000 to 9.000]
  Diarrhea: number analyzed (Participants) | 143 | 117
  Diarrhea | 6.000 [5.000 to 9.000] | 4.000 [3.000 to 6.000]
  Feeling hot or feverish: number analyzed (Participants) | 356 | 350
  Feeling hot or feverish | 3.000 [NA to NA] — Due to variability of data, the number of participants with events available was not sufficient for the calculation of the limits using Kaplan-Meier method. | 4.000 [3.000 to 4.000]
  Headache: number analyzed (Participants) | 429 | 424
  Headache | 5.000 [4.000 to 5.000] | 5.000 [5.000 to 6.000]
  Nausea: number analyzed (Participants) | 180 | 165
  Nausea | 4.000 [3.000 to 5.000] | 4.000 [3.000 to 5.000]
  Stuffy or runny nose: number analyzed (Participants) | 491 | 484
  Stuffy or runny nose | 5.000 [4.000 to 6.000] | 7.000 [6.000 to 7.000]
  Sore throat: number analyzed (Participants) | 371 | 381
  Sore throat | 4.000 [4.000 to 5.000] | 5.000 [4.000 to 6.000]
  Vomit: number analyzed (Participants) | 52 | 43
  Vomit | 3.000 [2.000 to 4.000] | 3.000 [2.000 to 7.000]

10. Secondary Outcome: Time to Sustained Resolution of Each COVID-19 Signs and Symptoms Through Day 28
Description: Sustained resolution was defined as when targeted symptoms are scored as absent for 4 consecutive days. The first day of the 4 consecutive-day period was considered the first event date. In this outcome measure time to sustained resolution is reported consolidated for each COVID-19 signs and symptoms.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants randomly assigned to study intervention, who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomized. Here ''Overall Number of Participants Analyzed''=participants evaluable for this outcome measure and ''number analyzed''= participants evaluable at specified time points.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 654 | 634
Days
  Muscle or body aches: number analyzed (Participants) | 466 | 449
  Muscle or body aches | 8.000 [7.000 to 9.000] | 9.000 [7.000 to 10.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 222 | 205
  Shortness of breath or difficulty breathing | 7.000 [5.000 to 7.000] | 8.000 [7.000 to 11.000]
  Chills or shivering: number analyzed (Participants) | 318 | 319
  Chills or shivering | 4.000 [3.000 to 5.000] | 5.000 [4.000 to 6.000]
  Cough: number analyzed (Participants) | 512 | 502
  Cough | 11.000 [10.000 to 12.000] | 12.000 [11.000 to 13.000]
  Diarrhea: number analyzed (Participants) | 143 | 117
  Diarrhea | 6.000 [6.000 to 8.000] | 5.000 [4.000 to 6.000]
  Feeling hot or feverish: number analyzed (Participants) | 356 | 350
  Feeling hot or feverish | 4.000 [3.000 to 5.000] | 5.000 [5.000 to 6.000]
  Headache: number analyzed (Participants) | 429 | 424
  Headache | 7.000 [7.000 to 9.000] | 9.000 [8.000 to 10.000]
  Nausea: number analyzed (Participants) | 180 | 165
  Nausea | 6.000 [4.000 to 7.000] | 5.000 [4.000 to 7.000]
  Stuffy or runny nose: number analyzed (Participants) | 491 | 484
  Stuffy or runny nose | 9.000 [7.000 to 10.000] | 10.000 [9.000 to 11.000]
  Sore throat: number analyzed (Participants) | 371 | 381
  Sore throat | 6.000 [6.000 to 7.000] | 8.000 [7.000 to 8.000]
  Vomit: number analyzed (Participants) | 52 | 43
  Vomit | 3.000 [2.000 to 4.000] | 3.000 [2.000 to 7.000]

11. Secondary Outcome: Percentage of Participants With Progression to Worsening Status of COVID-19 Signs and Symptoms
Description: Participants recorded a daily severity rating of their symptom severity over the past 24 hours based on a 4-point scale in which 0 was reported if no symptoms were present; 1 if mild; 2 if moderate; and 3 if severe. Vomiting and diarrhea was rated on a 4-point frequency scale where 0 is reported for no occurrence, 1 (mild) for 1 to 2 times, 2 (moderate) for 3 to 4 times, and 3 (severe) for 5 or greater. Progression to a worsening status for any targeted symptom was based up on increasing severity (i.e. the first time any targeted symptoms worsened after treatment relative to baseline).
Time Frame: From Day 1 to Day 28
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 648 | 633
Percentage of participants | 75.463 | 78.515
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo; Main effects of treatment, geographic region, symptom onset duration (<=3, >3), baseline SARS-CoV-2 serology status (positive/negative), vaccination status (complete/not vaccinated) and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL); Test type: Superiority; p = 0.1086, Regression, Logistic; Odds Ratio (OR) = 0.802, 95% CI 2-sided [0.613 to 1.050]

12. Secondary Outcome: Percentage of Participants With Resting Peripheral Oxygen Saturation Greater Than or Equal to (>=) 95% at Day 1 and Day 5
Description: Percentage of participants with a resting peripheral oxygen saturation >=95% were reported in this outcome measure.
Time Frame: Day 1 and Day 5
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 638 | 604
Percentage of participants
  Day 1: number analyzed (Participants) | 16 | 28
  Day 1 | 62.500 | 67.857
  Day 5 | 94.671 | 93.212
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg; Test type: Superiority; p = 0.3262, Breslow-Day Test; Odds Ratio (OR) = 50.333, 95% CI 2-sided [13.163 to 192.472]
Statistical Analysis 2: Comparison: Placebo; Odds ratio for Day 5 vs Day 1; Test type: Superiority; Odds Ratio (OR) = 22.224, 95% CI 2-sided [8.360 to 59.080]

13. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-07321332
Time Frame: Day 1: 1 hour post dose; Day 5: 0 minutes pre-dose
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received. A randomized but not treated participant was excluded from the safety analyses. Here ''Overall Number of Participants Analyzed''=participants evaluable for this outcome measure and ''number analyzed''= participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 287
Nanograms per milliliter
  Day 1 (1 hour post-dose): number analyzed (Participants) | 104
  Day 1 (1 hour post-dose) | 2437 (1791.3)
  Day 5 (0 minutes pre-dose) | 3468 (2454.7)

14. Secondary Outcome: Change From Baseline in Logarithm to Base10 (Log10) Transformed Viral Load at Days 3, 5, 10 and 14
Description: Nasal samples were collected to estimate the viral load in participants in terms of logarithm to base 10 (log10) copies per milliliter.
Time Frame: Baseline, Days 3, 5, 10 and 14
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Log 10 copies per milliliter
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 515 | 493
Log 10 copies per milliliter
  Day 3 | -2.302 (0.096) | -1.565 (0.098)
  Day 5: number analyzed (Participants) | 505 | 480
  Day 5 | -3.669 (0.090) | -2.835 (0.093)
  Day 10: number analyzed (Participants) | 489 | 478
  Day 10 | -4.873 (0.081) | -4.642 (0.082)
  Day 14: number analyzed (Participants) | 508 | 484
  Day 14 | -5.464 (0.072) | -5.249 (0.075)

ADVERSE EVENTS:
Time Frame: SAEs and Non-SAEs: From Day 1 to Week 24; All-cause mortality: till Week 24
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety population comprised of all participants who received at least 1 dose of study intervention during the study.
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/654 | 1/634
Serious Adverse Events (participants affected / at risk) | 8/654 | 13/634
Other Adverse Events (participants affected / at risk) | 120/654 | 71/634
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir 300 mg + Ritonavir 100 mg (N=654) | Placebo (N=634)
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 3 | 8
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia aspiration (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Osmotic demyelination syndrome (Nervous system disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir 300 mg + Ritonavir 100 mg (N=654) | Placebo (N=634)
Diarrhoea (Gastrointestinal disorders) | 26 | 19
Dyspepsia (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 21 | 17
Vomiting (Gastrointestinal disorders) | 11 | 11
Activated partial thromboplastin time prolonged (Investigations) | 7 | 12
Alanine aminotransferase increased (Investigations) | 14 | 8
Aspartate aminotransferase increased (Investigations) | 9 | 4
Blood thyroid stimulating hormone increased (Investigations) | 4 | 7
Fibrin D dimer increased (Investigations) | 8 | 9
Dysgeusia (Nervous system disorders) | 44 | 3
Headache (Nervous system disorders) | 6 | 9

LIMITATIONS AND CAVEATS:
In participant flow, there was discontinuations due to AE, which was captured under "Death" as reason for discontinuation. Adverse event was COVID-19 pneumonia and the participant died due to that event and discontinued study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT05011513/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05011513/SAP_001.pdf